CLINICAL TRIAL: NCT00006357
Title: Dose Finding and Phase II Study of STI 571 in Advanced Soft Tissue Sarcoma
Brief Title: STI571 in Treating Patients With Recurrent or Refractory Soft Tissue Sarcoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Purpose: Treatment
Other Study IDs: EORTC-62001-16003; EORTC-62001; EORTC-16003; NOVARTIS-CSTI5710203
Record Dates: First submitted 2000-10-04; First posted 2004-04-26 (Estimated); Last update posted 2012-09-24 (Estimated); Status verified 2012-09

CONDITIONS: Endometrial Cancer; Gastrointestinal Stromal Tumor; Ovarian Cancer; Sarcoma; Small Intestine Cancer
Keywords: adult angiosarcoma; adult fibrosarcoma; adult leiomyosarcoma; adult liposarcoma; adult neurofibrosarcoma; adult synovial sarcoma; recurrent adult soft tissue sarcoma; small intestine leiomyosarcoma; adult alveolar soft-part sarcoma; adult epithelioid sarcoma; adult malignant fibrous histiocytoma; adult malignant hemangiopericytoma; adult malignant mesenchymoma; adult rhabdomyosarcoma; ovarian stromal cancer; recurrent uterine sarcoma; uterine carcinosarcoma; uterine leiomyosarcoma; endometrial stromal sarcoma; ovarian sarcoma; gastrointestinal stromal tumor
MeSH Terms: conditions — Endometrial Neoplasms; Gastrointestinal Stromal Tumors; Ovarian Neoplasms; Sarcoma; Hemangiosarcoma; Fibrosarcoma; Leiomyosarcoma; Liposarcoma; Neurofibrosarcoma; Sarcoma, Synovial; Sarcoma, Alveolar Soft Part; Histiocytoma, Malignant Fibrous; Hemangiopericytoma, Malignant; Malignant mesenchymal tumor; Rhabdomyosarcoma; Sarcoma, Endometrial Stromal | interventions — Imatinib Mesylate

INTERVENTIONS:
Drug: imatinib mesylate

SUMMARY:
RATIONALE: STI571 may interfere with the growth of cancer cells and may be an effective treatment for soft tissue sarcoma.

PURPOSE: Phase I/II trial to study the effectiveness of STI571 in treating patients who have recurrent or refractory soft tissue sarcoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the maximum tolerated dose and associated toxicity of STI571 in patients with refractory or recurrent soft tissue sarcoma. II. Determine the pharmacokinetic profile of this treatment regimen in these patients. III. Determine the objective response and duration of response in these patients with this treatment regimen.

OUTLINE: This is a dose escalation and dose efficacy, multicenter study. In the dose efficacy portion, patients are stratified according to disease type (gastrointestinal stromal tumor vs all other soft tissue sarcomas). Phase I: Patients receive oral STI571 daily for a maximum of 24 months in the absence of disease progression or unacceptable toxicity. Cohorts of 3-8 patients receive escalating doses of STI571 until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose at which 2 of 6-8 patients experience dose limiting toxicities. The recommended phase II dose is defined as the dose preceding the MTD. Phase II: Patients receive the recommended phase II dose of STI571 as in phase I. Patients are followed every 8 weeks until disease progression, and then every 16 weeks thereafter.

PROJECTED ACCRUAL: Approximately 47-72 patients (7-32 in phase I and 40 in phase II) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed soft tissue sarcoma Malignant fibrous histiocytoma Liposarcoma Rhabdomyosarcoma Synovial sarcoma Malignant paraganglioma Fibrosarcoma Leiomyosarcoma Angiosarcoma Hemangiopericytoma Neurogenic sarcoma Unclassified sarcoma Miscellaneous sarcoma (including mixed mesodermal tumors of the uterus) Gastrointestinal stromal tumor (GIST) (must be c-kit positive) No malignant mesothelioma, chondrosarcoma, neuroblastoma, osteosarcoma, Ewing's sarcoma, or embryonal rhabdomyosarcoma Phase I study and nonGIST phase II study patients: Must have received one prior first line combination chemotherapy regimen or two first line single agent regimens Adjuvant chemotherapy not considered first line, unless disease progression within 6 months of treatment Phase II GIST patients: No more than one prior first line combination chemotherapy regimen or two first line single agent regimens Adjuvant chemotherapy not considered first line, unless disease progression within 6 months of treatment Measurable disease with evidence of progression in past 6 weeks Osseous lesions and pleural effusions not considered measurable No symptomatic or known CNS metastases

PATIENT CHARACTERISTICS: Age: 15 and over Performance status: WHO 0-1 Life expectancy: Not specified Hematopoietic: Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 1.8 mg/dL Albumin at least 25 g/L Renal: Creatinine no greater than 1.4 mg/dL OR Creatinine clearance greater than 65 mL/min Cardiovascular: No history of cardiovascular disease Other: No prior or concurrent second primary malignant tumors except adequately treated carcinoma in situ of the cervix or basal cell carcinoma No other severe illness (including psychosis) Not pregnant Fertile patients must use effective contraception during and for 6 months following study

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics At least 4 weeks since prior chemotherapy No other concurrent local or systemic chemotherapy Endocrine therapy: No concurrent systemic corticosteroid therapy Radiotherapy: No prior radiotherapy to sole index lesion Concurrent radiotherapy to any lesion allowed if not the sole target lesion Surgery: Not specified Other: No prior embolization to sole index lesion No other concurrent investigational drug No concurrent warfarin

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2000-08; Primary Completion 2001-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacob Verweij, MD, PhD, Study Chair — Daniel Den Hoed Cancer Center at Erasmus Medical Center
Locations (16):
- Belgium (2):
  - Universitair Ziekenhuis Antwerpen, Edegem
  - U.Z. Gasthuisberg, Leuven
- Denmark (3):
  - Aarhus Kommunehospital, Aarhus
  - Rigshospitalet, Copenhagen
  - Herlev Hospital - University Hospital of Copenhagen, Herlev
- France (2):
  - Centre Leon Berard, Lyon
  - Institut Gustave Roussy, Villejuif
- Netherlands (5):
  - Antoni van Leeuwenhoekhuis, Amsterdam
  - Academisch Ziekenhuis Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen
  - Rotterdam Cancer Institute, Rotterdam
- United Kingdom (4):
  - Royal Marsden NHS Trust, London, England
  - Christie Hospital N.H.S. Trust, Manchester, England
  - Nottingham City Hospital NHS Trust, Nottingham, England
  - Weston Park Hospital, Sheffield, England

REFERENCES:
- [Result] van Erp N, Gelderblom H, van Glabbeke M, Van Oosterom A, Verweij J, Guchelaar HJ, Debiec-Rychter M, Peng B, Blay JY, Judson I. Effect of cigarette smoking on imatinib in patients in the soft tissue and bone sarcoma group of the EORTC. Clin Cancer Res. 2008 Dec 15;14(24):8308-13. doi: 10.1158/1078-0432.CCR-08-1303. PMID 19088049
- [Result] Judson I, Ma P, Peng B, Verweij J, Racine A, di Paola ED, van Glabbeke M, Dimitrijevic S, Scurr M, Dumez H, van Oosterom A. Imatinib pharmacokinetics in patients with gastrointestinal stromal tumour: a retrospective population pharmacokinetic study over time. EORTC Soft Tissue and Bone Sarcoma Group. Cancer Chemother Pharmacol. 2005 Apr;55(4):379-386. doi: 10.1007/s00280-004-0876-0. Epub 2004 Dec 9. PMID 15592836
- [Result] Debiec-Rychter M, Dumez H, Judson I, Wasag B, Verweij J, Brown M, Dimitrijevic S, Sciot R, Stul M, Vranck H, Scurr M, Hagemeijer A, van Glabbeke M, van Oosterom AT; EORTC Soft Tissue and Bone Sarcoma Group. Use of c-KIT/PDGFRA mutational analysis to predict the clinical response to imatinib in patients with advanced gastrointestinal stromal tumours entered on phase I and II studies of the EORTC Soft Tissue and Bone Sarcoma Group. Eur J Cancer. 2004 Mar;40(5):689-95. doi: 10.1016/j.ejca.2003.11.025. PMID 15010069
- [Result] Verweij J, van Oosterom A, Blay JY, Judson I, Rodenhuis S, van der Graaf W, Radford J, Le Cesne A, Hogendoorn PC, di Paola ED, Brown M, Nielsen OS. Imatinib mesylate (STI-571 Glivec, Gleevec) is an active agent for gastrointestinal stromal tumours, but does not yield responses in other soft-tissue sarcomas that are unselected for a molecular target. Results from an EORTC Soft Tissue and Bone Sarcoma Group phase II study. Eur J Cancer. 2003 Sep;39(14):2006-11. PMID 12957454
- [Result] van Oosterom AT, Judson IR, Verweij J, Stroobants S, Dumez H, Donato di Paola E, Sciot R, Van Glabbeke M, Dimitrijevic S, Nielsen OS; European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. Update of phase I study of imatinib (STI571) in advanced soft tissue sarcomas and gastrointestinal stromal tumors: a report of the EORTC Soft Tissue and Bone Sarcoma Group. Eur J Cancer. 2002 Sep;38 Suppl 5:S83-7. doi: 10.1016/s0959-8049(02)80608-6. PMID 12528778
- [Result] van Oosterom AT, Judson I, Verweij J, Stroobants S, Donato di Paola E, Dimitrijevic S, Martens M, Webb A, Sciot R, Van Glabbeke M, Silberman S, Nielsen OS; European Organisation for Research and Treatment of Cancer Soft Tissue and Bone Sarcoma Group. Safety and efficacy of imatinib (STI571) in metastatic gastrointestinal stromal tumours: a phase I study. Lancet. 2001 Oct 27;358(9291):1421-3. doi: 10.1016/s0140-6736(01)06535-7. PMID 11705489